CLINICAL TRIAL: NCT03629951
Title: An Observational Study for Schizophrenia Relapse Prediction
Brief Title: A Study for Schizophrenia Relapse Prediction
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108481; NOPRODSCH4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-07-25; First posted 2018-08-14 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Antipsychotic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Schizophrenia: Participants will not receive any intervention as a part of this study. Participants with a diagnosis of schizophrenia or schizoaffective disorder receiving oral antipsychotics (OAP) for example, risperidone (1 to 6 milligram [mg] once daily [OD] to twice a day [BID]), olanzapine (5 to 20 mg OD), haloperidol (5 to 20 mg OD to thrice a day [TID]) etc, per their treating physician/clinician instruction will be observed. The primary data source for this study will be the clinical assessments by the treating physician of each participant conducted as a part of routine clinical practice.
  Interventions: Drug: Oral Antipsychotics (OAP)

INTERVENTIONS:
Drug: Oral Antipsychotics (OAP) — This is an observational study. Participants enrolled in this study will continue to receive routine treatment of OAPs for example, risperidone (1 to 6 mg OD to BID), olanzapine (5 to 20 mg OD), haloperidol (5 to 20 mg OD to TID) etc, as directed by their treating physician.

SUMMARY:
The purpose of this study is to identify if there are self-reported/caregiver reported or objective measures that can predict near-term relapse (within 1 month or at another identified time point before meeting the criteria for relapse) or early symptomatic changes indicative of pre-relapse.

ELIGIBILITY:
Inclusion Criteria:

* Participants and their legally acceptable representative where applicable must be able to sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate for the duration of the study
* Have a clinical diagnosis of schizophrenia made by a clinician with understanding of the criteria for schizophrenia or schizoaffective disorder, per the Diagnostic and Statistical Manual of Mental Disorders - 5th edition (DSM-5), and had at least 1 relapse, in the opinion of the investigator, within the last 12 months prior to date of informed consent
* Must be receiving an OAP treatment regimen at the time of enrollment
* Must be able to speak, read, and understand English and/or the local Indian language as the patient reported outcome instruments will be validated in regional languages
* Caregivers/Informants should be able to sign an ICF indicating that he or she understands the purpose of and procedures required for the study and is willing to participate for the duration of the study

Exclusion Criteria:

* Has treatment resistant schizophrenia (that is, currently receiving clozapine or electroconvulsive therapy [ECT])
* Is on long-acting injectable antipsychotic regimen at the time of screening
* Has a moderate to severe substance use disorder (other than nicotine), as determined by the investigator
* Has a significant risk of suicide or active suicidality with a plan as indicated by the Columbia-Suicide Severity Rating Scale (C-SSRS) assessment
* Has an immediate need for hospitalization (that is, the participant is already in a relapse)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants with clinical diagnosis of schizophrenia receiving an oral antipsychotic (OAP) treatment regimen directed by their treating clinician will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Relapse | Up to Approximately 3 years
  Relapse is defined as achieving any of the following: clinically meaningful worsening of symptoms as determined by the treating physician's judgment; involuntary or voluntary admission to a psychiatric hospital for decompensation of the participant's schizophrenic symptoms (psychiatric hospitalization); deliberate self-injury and/or violent behavior resulting in clinically significant injury to the participant or another person or property damage; suicidal or homicidal ideation and aggressive behavior considered as clinically significant (in frequency and severity) in the treating physician's judgment; an increase of at least 2 points from the lowest reported Clinical Global Impression-Severity (CGI-S) score (ranging from 1 [not ill] to 7 [extremely severe]) captured either at baseline or post baseline. Number of participants with relapse will be determined.

SECONDARY OUTCOMES:
Number of Participants in each Clinical State of Schizophrenia | Up to approximately 3 years
  Number of participants in each clinical state (Acute, Stable, and Remission) of schizophrenia will be assessed. The clinical states are defined as: 'Acute' - Clinical Global Impression-Severity (CGI-S) score (ranging from 1 [not ill] to 7 [extremely severe]) greater than or equal to (>=)5 anytime during the study; 'Stable' (Tier I) - control of acute symptoms, defined as having a CGI-S score of less than or equal to (<=)3 for a minimum of 3 months and/or (Tier II) - stable dosage of oral antipsychotic (OAPs) for a minimum of 3 months and control of acute symptoms, defined as having a CGI-S score of <=4 for a minimum of 3 months; and 'Remission' - a continuous CGI-S scale score of <=2 for 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- India (10):
  - Panchshil Hospital, Ahmedabad
  - Ratandeep Multispeciality Hospital, Ahmedabad
  - Asha hospital, Hyderabad
  - Mahendru Psychiatric Centre, Kanpur
  - Ahana Hospitals, Madurai
  - Kasturba Medical College Hospital, Manipal
  - Meera Hospital, Mumbai
  - Meditrina Institute of Medical Sciences, Nagpur
  - GMERS Medical College and Hospital, Vadodara
  - Deva Institute of Health Care and Research Pvt Ltd, Varanasi